CLINICAL TRIAL: NCT03587246
Title: Comparison of Uterine Peristaltic Wave Frequencies Between Pregnant and Non-pregnant Women in Embryo Transfer Cycles
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Kamolrat Daoudom, Doctor, Chulalongkorn University
Other Study IDs: 375/61
Record Dates: First submitted 2018-07-02; First posted 2018-07-16 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Uterine Peristaltic Frequencies Between Pregnant and Non-pregnant Women in Embryo Transfer Cycles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood collection for estradiol progesterone LH FSH level
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women
  Interventions: Diagnostic Test: 3DTVUS : Uterine peristaltic frequencies
- non-pregnant women
  Interventions: Diagnostic Test: 3DTVUS : Uterine peristaltic frequencies

INTERVENTIONS:
Diagnostic Test: 3DTVUS : Uterine peristaltic frequencies — Perform three-dimensional transvaginal ultrasonography To observe uterine peristaltic frequencies in embryo transfer cycles

SUMMARY:
Eligibility criteria

* Infertile woemn undergo IVF & embryo transfer cycles at infertility clinic at King Chulalongkorn Memorial Hospital Measurement
* Uterine peristaltic wave frequencies & Junctional zone thickness by 3D-TVUS on the day of oocyte retrieval in fresh embryo transfer participants & day before progesterone supplementation in frozen-thawed embryo transfer participants
* Serum progesterone & estradiol level in the same day

DETAILED DESCRIPTION:
The patients who were planning to undergo fresh embryo transfer cycles used GnRH antogonist protocol. Ovarian stimulation was initiated on the menstrual cycle day 3 with use of daily subcutaneous injection of gonodotrophin; human menopausal gonadotrophin (Menopur®), recombinant FSH-alpha (Gonal-F®), recombinant FSH-beta (Puregon®). After 5 days of stimulation, the dosage of gonadotrophin was adjusted based on ovarian response, as assessed by follicular size monitoring and serum estradiol levels. To prevent premature LH surges, ganirelix (Orgalutran®) was administered by subcutaneous injection when at least one follicle reached a diameter of 13 mm. When the leading follicle reached 18 mm in diameter, final oocyte maturation was triggered by subcutaneous injection of recombinant hCG (Ovidrel®) 0.25 mg or double triggered by addition subcutaneous injection of triptorelin (Diphereline®) 0.1 mg. Oocyte retrieval was performed 36 hours after drug administration. Insemination of retrieved oocytes was performed by intracytoplasmic sperm injection (ICSI). Progesterone supplement was started on the day of ovum pickup with 400 mg-micronized vaginal progesterone pessary (Cyclogest®) two times a day. Embryo transfer was performed on day 4 to day 6 of progesterone supplement.

The patients who were planning to undergo frozen embryo transfer cycles used artificial endometrial preparation or natural cycles. Endometrial priming was achieved with daily oral estradiol valerate (Progynova®) 6-8 mg per day beginning on the

￼cycle day 3 for 12 days. Endometrial thickness was assessed by transvaginal ultrasonography. Once the endometrium thickness reaches 8 mm with trilaminar appearance, 400-mg micronized vaginal progesterone pessary was started daily. Embryo transfer was performed on day 4 to day 6 of progesterone supplement. In the participants were not achieved the goal, dosage of oral estradiol valerate was increased and/or 50 microgram-transdermal estradiol hemihydrates (Climara®) was added. Two to three days after adjusted dose, the endometrial thickness was reassessed and progesterone was administered as mentioned above if the goal was reached. Cycle cancellation was chosen if the thickness was not optimal.

Embryo transfer was performed following ASRM guidance using either soft or metallic catheter. The procedure was done gently avoiding fundal contact with transabdominal ultrasonography monitoring.

￼All participants were examined uterine peristaltic wave frequencies and thickness of junctional zone two times by three- dimensional transvaginal ultrasonography (3D-TVUS). The first measurement was performed on day 2 of menstrual cycle. The second measurement was performed on the day planning to start progesterone administration in frozen-thawed embryo transfer protocol and the day of oocyte retrieval in fresh embryo transfer protocol.

Three-dimensional ultrasonography machine, Voluson S6 (GE, USA), was used with RIC5-9W real-time 4D micro-convex endovaginal curved linear probe by single operator. All participants were instructed to avoid sexual activity before evaluation for two days. The patient was lying relaxed in a lithotomy position after emptying the bladder. To avoid stimulating the cervix, the probe was gently introduced into the vagina and uterine peristaltic wave was measured first. Two-minute video of fixed mid-sagittal plane of uterus was recorded. Three dimensional sonographic features were obtained by applying volume box covered the mid-sagittal plane of uterus. Coronal plane of uterus was appeared after automatic sweep of mechanical transducer by multiplanar and OMNI view. Speckle reduction imaging (SRI) and volume contrast imaging (VCI) modality was set up at SRI 0-2 and VCI 2-4 mm. Thickness of junctional zone was measured as the distance from the basal endometrium to the internal layer of the outer myometrium, which appeared as relative hypoechoic linear lining around the endometrium. All sides of uterine wall were evaluated; fundal, lateral, anterior, and posterior wall. Each side was measured at two regions, the thickest and the thinnest distance and the average thickness of each wall was obtained by dividing of the sum of thickest and thinnest area. Finally, the average thickness of four uterine walls was obtained. Uterine peristaltic wave frequencies were analyzed with 4X of regular speed using a VLC media player by two independent observers. The mean of

￼peristaltic wave frequencies between two persons were obtained if the frequencies were not concordance.

Hormonal levels were checked for analysis two times in each patient. First measurement, serum luteinizing hormone (LH) and estradiol hormone levels were measured at day 2 of menstrual cycle in all participants. The patients in fresh embryo transfer cycles, serum follicle stimulating hormone (FSH) measurement was added. Second measurement, serum estradiol and progesterone hormone levels were checked in the same day of 3D-TVUS assessment.

Two weeks after embryo transfer, serum beta-hCG was first measured. In the patients with rising hCG level, serum level was reassessed at week 3 and week 4 after embryo transfer and transvaginal ultrasonography was performed at week 4 after the transfer. Vaginal progesterone was continued in the same dose and intramuscular 17-hydroxyprogesterone caproate (Depot- proluton®) was added weekly. Luteal support was continued until 12 weeks of gestation. In non-pregnant women, vaginal progesterone was stopped after first measurement of serum beta-hCG. Clinical pregnancy was defined as the presence of intrauterine gestational sac four weeks after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* women age < 45years
* BMI < 35 kg/m2
* at least one of good quality embryo in embryo transfer cycle by Istanbul consensus workshop morphologic grading Day3 : Grade 1-2, Day4 : Grade 1-2 , Day5 : stage of development grade 2-4

Exclusion Criteria:

* structural intrauterine cavity distortion
* leiomyoma FIGO subclassification 3
* adenomyosis
* recurrent pregnancy loss
* recurrent implantation failure
* urerine relaxant drugs
* difficult embryo transfer

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Infertile women undergone IVF cycle treatments and embryo transfer cycles in infertile clinic at King Chulalongkorn Memorial hospital from 2018-2019
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Association of uterine peristaltic frequencies with pregnancy outcomes of embryo transfer cycles | 3 minutes
  For frozen-thawed embryo cycles : observation on the day of 8 mm-triple layer endometrial thickness For fresh embryo transfer cycles : observation on the day of oocyte retrieval procedure

SECONDARY OUTCOMES:
Association of junctional zone thickness with pregnancy outcomes in embryo transfer cycles | 3 minutes
  For frozen-thawed embryo cycles : observation on the day of 8 mm-triple layer endometrial thickness For fresh embryo transfer cycles : observation on the day of oocyte retrieval procedure
Association of uterine peristaltic frequencies and junctional zone thickness between fresh embryo transfer cycles & frozen-thawed embryo transfer cycles | 3 minutes
  For frozen-thawed embryo cycles : observation on the day of 8 mm-triple layer endometrial thickness For fresh embryo transfer cycles : observation on the day of oocyte retrieval procedure
Association of uterine peristaltic frequencies with junctional zone thickness | 3minutes
  For frozen-thawed embryo cycles : observation on the day of 8 mm-triple layer endometrial thickness For fresh embryo transfer cycles : observation on the day of oocyte retrieval procedure

CONTACTS AND LOCATIONS:
Overall Officials: KamolratD Daoudom, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No